CLINICAL TRIAL: NCT02530125
Title: Phase II Study of Pidilizumab (MDV9300) in Patients With Diffuse Large B-Cell Lymphoma Following First Remission
Brief Title: Pidilizumab in Treating Patients With Stage III-IV Diffuse Large B-Cell Lymphoma Following First Remission
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: sponsor decided to discontinue development of the study drug.
Sponsor: Northwestern University (Other)
Collaborators: Gateway for Cancer Research (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jane N. Winter, Principal Investigator, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 15H08; NCI-2015-01415 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STU00200695; NU 15H08 (Other: Northwestern University); P30CA060553 (NIH)
Record Dates: First submitted 2015-08-19; First posted 2015-08-20 (Estimated); Results first posted 2018-03-19 (Actual); Last update posted 2018-03-19 (Actual); Status verified 2017-04

CONDITIONS: Stage III Diffuse Large B-Cell Lymphoma; Stage IV Diffuse Large B-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — pidilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (pidilizumab) (Experimental): Patients receive pidilizumab IV over approximately 5 hours on day 1. Treatment repeats every 42 days for 3 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Biological: Pidilizumab

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Pidilizumab — Given IV
  Other Names: CT-011

SUMMARY:
The purpose of this study is to evaluate pidilizumab and its effect, bad and/or good, on the immune system in relation to its ability to fight cancer cells. Many cancers can be brought to a phase called complete remission (no cancer is found) but have a chance that they may come back. Researchers are working to improve therapy and to find new drugs that lower the chance of disease coming back. This study uses a drug called pidilizumab. The drug targets our immune system. It can change how our immune system finds cancer cells. The drug may kill any remaining cancer cells that we cannot see with computed tomography (CT) scans. The drug, pidilizumab, is being studied in other cancers.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the rate of response, whereby either cluster of differentiation (CD)4+CD25+programmed death 1 ligand 1 (PD-L1)+ T lymphocytes or CD4+CD62L+CD127+ T lymphocytes has an "increase" following administration of pidilizumab in patients with diffuse large B-cell lymphoma (DLBCL) that have completed induction chemotherapy.

SECONDARY OBJECTIVES:

I. To determine the toxicity and tolerability of pidilizumab therapy following induction chemotherapy.

II. To estimate the progression free survival (PFS) at 2 years. III. To estimate the overall survival (OS) at 2 years. IV. To estimate time to second line chemotherapy (TSLC) at 2 years.

TERTIARY OBJECTIVES:

I. To characterize programmed death 1 (PD-1) pathway specific expression markers from the diagnostic biopsy specimens.

II. To characterize serum biomarkers of immune and inflammatory response during treatment with pidilizumab.

III. To characterize levels of soluble PD-L1 related to treatment with pidilizumab.

OUTLINE:

Patients receive pidilizumab intravenously (IV) over approximately 5 hours on day 1. Treatment repeats every 42 days for 3 courses in the absence of disease progression or unacceptable toxicity.

After completion of treatment, patients are followed up at 30 days and then every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed de novo DLBCL by the 4th edition of the World Health Organization (WHO) Classification of Tumors of Hematopoietic and Lymphoid Tissues published in 2008; patients with transform lymphoma are excluded; patients with known primary mediastinal large B-cell lymphoma (PMLBCL) are excluded; patients with known c-v-myc avian myelocytomatosis viral oncogene homolog (c-myc) translocation (by fluorescence in situ hybridization) positive DLBCL are eligible for enrollment; c-myc testing prior to study enrollment is not required; availability of diagnostic biopsy samples in encouraged for the exploratory analysis but not required for enrollment; patients with "double-hit" or "triple-hit" lymphoma are eligible for enrollment
* Previously completed anthracycline-based induction chemotherapy with standard regimens including rituximab, cyclophosphamide, doxorubicin hydrochloride, vincristine sulfate, and prednisone (R-CHOP), dose adjusted (DA)-etoposide, prednisone, vincristine sulfate, doxorubicin hydrochloride, cyclophosphamide (EPOCH), and rituximab (R), and R-hyper cyclophosphamide, vincristine sulfate, doxorubicin hydrochloride, dexamethasone, methotrexate, and cytarabine (CVAD); patients need a minimum of 6 cycles of treatment; initial treatment with pidilizumab must be administered between 30-90 days from last dose of induction chemotherapy
* Complete remission (CR) according to the Revised Response Criteria for Malignant Lymphoma after first-line treatment

  * Diagnostic CT scans with contrast of chest, abdomen, and pelvis must have been performed within 8 weeks from the first day of the last cycle of R-chemotherapy; a neck CT will be required if the patient had involvement of the neck region at initial diagnosis
  * A negative fludeoxyglucose F 18 (FDG)-positron emission tomography (PET)/CT scan performed within 8 weeks from the first day of the last cycle of R-chemotherapy and confirming CR, with negative defined as a score of 1-3 on the Deauville 5-point scale used to quantify radionucleotide density in PET scans as determined locally; PET positive/indeterminate lesions which are confirmed on biopsy to harbor no active lymphoma will be considered negative for determination of CR status
  * If positive bone marrow involvement at initial diagnosis the patient must have a negative bone marrow biopsy following R-chemotherapy to confirm the CR
* Stage III/IV disease by Ann Arbor Staging
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Any National Comprehensive Cancer Network (NCCN)-International Prognostic Index (IPI) score; a calculated score required for enrollment
* Absolute neutrophil count (ANC) >= 1000
* Platelet count >= 50,000
* Total bilirubin =< 2 x upper limit of normal (ULN) or if total bilirubin is > 2 x ULN, the direct bilirubin must be normal
* Alkaline (Alk.) phosphatase =< 3 x ULN
* Aspartate aminotransferase (AST) =< 3 x ULN
* Creatinine =< 2 x ULN or creatinine clearance (CrCl) > 30 ml/min
* Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test at enrollment; FCBP must either commit to abstinence from heterosexual intercourse or commit to the use of 2 acceptable methods of birth control; a FCBP is any woman, regardless of sexual orientation or whether they have undergone tubal ligation, who meets the following criteria: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months)
* Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy
* All subjects must have given signed, informed consent prior to registration on study

Exclusion Criteria:

* Active malignancy requiring therapy such as radiation, chemotherapy, or immunotherapy; exceptions to this are as follows: localized nonmelanotic skin cancer and any cancer that in the judgment of the investigator has been treated with curative intent and will not interfere with the study treatment plan and response assessment
* Known central nervous system (CNS) involvement
* Prior stem cell transplantation (autologous or allogeneic)
* Persistent diarrhea or malabsorption > National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) grade 2, despite medical management
* Subjects with known immunodeficiency, known autoimmune disease, or concurrent use of immunomodulatory agents
* Any cancer directed therapies between completion of induction chemotherapy and treatment on protocol
* Known hypersensitivity to murine or chimeric antibodies or proteins
* Presence of co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens; this includes, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Subjects with known human immunodeficiency virus (HIV) infection
* Subjects with known active hepatitis B virus (HBV) and hepatitis C virus (HCV) infection
* Women must not be pregnant or breast-feeding
* Unwillingness or inability to comply with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jane Winter, MD, Principal Investigator — Northwestern University
Locations (2):
- United States (2):
  - Georgia Regents University Medical Center, Augusta, Georgia
  - Northwestern University, Chicago, Illinois

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened for accrual on August 4, 2016 with an accrual goal of up to 30 patients. The manufacturer of pidilizumab requested accrual be suspended on November 15, 2016 and the study was permanently closed to accrual. The manufacturer discontinued pidilizumab due to issues with supply. 4 patients were registered and treated with pidilizumab.
Period: Completed Treatment
Arm/Group | Treatment (Pidilizumab)
Started | 4
Completed | 3
Not Completed | 1
Not completed — Early termination of study | 1
Period: Followed for Survival for 2 Years
Arm/Group | Treatment (Pidilizumab)
Started | 3
Completed | 0
Not Completed | 3
Not completed — Early termination of study | 3

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Pidilizumab)
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Response to Pidilizumab
Description: Response will be defined as the proportion of CD4+CD25+PD-L1+ T lymphocytes and CD4+CD62L+CD127+ T lymphocytes responders. Responders are defined as either a) a 50% increase or b) a half standard deviation increase in lymphocyte subsets. Lymphocyte subsets will be evaluated by flow cytometry on peripheral blood obtained at specified time points through the treatment period.
Time Frame: Baseline to up to 127 days. Study terminated before this timeframe. As a result insufficient data was collected to be analyzed.
Population: Study terminated early due to manufacturer decision to discontinue pidilizumab. As a result insufficient data was collected to be analyzed.
Arm/Group | Treatment (Pidilizumab)
Number analyzed (Participants) | 0

2. Secondary Outcome: The Frequency and Severity of Toxicity - Number of Grade 1, 2, 3, 4, and 5, Adverse Events Experienced During Treatment of Pidilizumab Defined by NCI CTCAE v 4.03.
Description: Adverse events (AEs) were graded according to the National Cancer Institute's Common Toxicity Criteria for Adverse Events (CTCAE) version 3.0. In general, AEs are graded according to the following:
  Grade 1 Mild AE Grade 2 Moderate AE Grade 3 Severe AE Grade 4 Life-threatening or disabling AE Grade 5 Death related to AE
Time Frame: Start of treatment, and at days 22, 43, 85, 127 and every 3 months for up to 2 years. Due to early termination of the study, AEs for all patients were collected throughout treatment and up to the point of termination of the study.
Population: This is only based of of 4 patients that received treatment of pidilizumab. Study terminated early due to manufacturer decision to discontinue pidilizumab.
Measure: Number; unit: Adverse events
Arm/Group | Treatment (Pidilizumab)
Number analyzed (Participants) | 4
Adverse events
  Grade 1 | 55
  Grade 2 | 10
  Grade 3 | 2
  Grade 4 | 0
  Grade 5 | 0

3. Secondary Outcome: Overall Survival (OS)
Description: To estimate the overall survival (OS) at 2 years
Time Frame: From study enrollment until death, or until last contact, assessed up to 2 years. Study terminated before this timeframe. As a result insufficient data was collected to be analyzed.
Population: as for outcome 1
Arm/Group | Treatment (Pidilizumab)
Number analyzed (Participants) | 0

4. Secondary Outcome: Progression Free Survival (PFS)
Description: To estimate the progression free survival (PFS) at 2 years. PFS will be defined as time from study enrollment until the first occurrence of disease relapse, progression, re-initiation of cytotoxic chemotherapy, or death due to disease, or until last contact if the patient did not experience any of these.
Time Frame: Up to 2 years. Study terminated before this timeframe. As a result insufficient data was collected to be analyzed.
Population: as for outcome 1
Arm/Group | Treatment (Pidilizumab)
Number analyzed (Participants) | 0

5. Secondary Outcome: Relapsed Disease
Time Frame: Up to 2 years. Study terminated before this timeframe. As a result insufficient data was collected to be analyzed.
Population: as for outcome 1
Arm/Group | Treatment (Pidilizumab)
Number analyzed (Participants) | 0

6. Secondary Outcome: Time to Second Line Chemotherapy (TSLC)
Description: To estimate time to second line chemotherapy (TSLC) at 2 years
Time Frame: Up to 2 years
Population: as for outcome 1
Arm/Group | Treatment (Pidilizumab)
Number analyzed (Participants) | 0

7. Other Pre Specified Outcome: Change in Soluble PD-L1 Levels
Description: Peripheral blood obtained at day 1 and day 127 will be analyzed and levels will be compared to evaluate for a change (increase/decrease) following treatment with pidilizumab.
Time Frame: as for outcome 1
Population: as for outcome 1
Arm/Group | Treatment (Pidilizumab)
Number analyzed (Participants) | 0

8. Other Pre Specified Outcome: Levels of Serum Biomarkers of Immune and Inflammatory Response
Description: Peripheral blood will be tested for serum levels of TNF-α, IFN-γ, IL-2, IL- 7, IL-9, and galectin-1. Levels will be compared from specified time points through treatment.
Time Frame: as for outcome 1
Population: as for outcome 1
Arm/Group | Treatment (Pidilizumab)
Number analyzed (Participants) | 0

9. Other Pre Specified Outcome: PD-1 and PD-L1 Pathway Specific Expression Markers
Description: Tissue sample slides from the diagnostic biopsy will be evaluated by immunohistochemistry for expression of PD-1 and PD-L1. Presence/absence (binary) of PD-1 and PD-L1 will be correlated with response to pidilizumab and clinical outcomes.
Time Frame: as for outcome 1
Population: as for outcome 1
Arm/Group | Treatment (Pidilizumab)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected over 1 year, 4 months [Time frame: Start treatment through 127 days and then every 3 months up to 2 years]
Description: The study was designed to collect adverse events at the following timepoints: Start of treatment, and at days 22, 43, 85, 127 and every 3 months for up to 2 years. Due to early termination of the study, AEs for all patients were collected throughout treatment and up until the point of termination of the study.
Arm/Group | Treatment (Pidilizumab)
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 1/4
Other Adverse Events (participants affected / at risk) | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Pidilizumab) (N=4)
Basal cell carcinoma (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Pidilizumab) (N=4)
Anemia (Blood and lymphatic system disorders) | 2 (3)
Constipation (Gastrointestinal disorders) | 2 (4)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 2 (2)
Edema limbs (General disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Neutrophil count decrease (Investigations) | 2 (2)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 3 (8)
Platelet count decreased (Investigations) | 2 (3)
White blood cell decreased (Investigations) | 2 (7)
Bronchial infection (Infections and infestations) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (7)
Hyperalbuminemia (Metabolism and nutrition disorders) | 2 (4)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2)
Oliguria (Renal and urinary disorders) | 1 (1)
Post nasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Hypertension (Vascular disorders) | 1 (2)
Hematoma (Vascular disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Study terminated early due to manufacturer decision to discontinue pidilizumab. As a result insufficient data was collected to be analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes